CLINICAL TRIAL: NCT01129349
Title: A Phase 1, Open-label, Dose Escalation Study of Oprozomib Administered Orally in Patients With Advanced Refractory or Recurrent Solid Tumors
Brief Title: Phase 1 Study of Oprozomib Administered Orally in Patients With Advanced Refractory or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-003
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Solid Tumors
Keywords: Solid Tumors
MeSH Terms: interventions — ONX 0912

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oprozomib (Experimental): Phase I, Dose Escalation, Single Arm, Open Label
  Interventions: Drug: Oprozomib

INTERVENTIONS:
Drug: Oprozomib — Oral administration of Oprozomib on Days 1-5 of a 14 day cycle

SUMMARY:
To evaluate the safety and tolerability of Oprozomib in patients with advanced refractory or recurrent solid tumors including determination of its Dose Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD) To determine the pharmacokinetics (PK) of Oprozomib To explore the anti-tumor activity of Oprozomib in this patient population including the overall response rate (ORR), the duration of responses (DOR), the progression-free survival (PFS) and time to progression (TTP) To define the pharmacodynamics (PDn) of Oprozomib.

DETAILED DESCRIPTION:
This is a Phase 1, open label, dose-escalation study to determine the safety, MTD, and PK/PDn of Oprozomib when administered orally (PO) on Days 1, 2, 3, 4, and 5 of a 14 day cycle in patients with advanced refractory or recurrent solid tumor malignancies for which standard curative measures do not exist or are no longer effective.

ELIGIBILITY:
Inclusion Criteria:

* Disease Related

  * Histologically confirmed advanced solid tumor that is refractory or recurrent after standard treatments.
  * At least one site of radiographically measurable disease of ≥ 2 cm in the largest dimension by traditional computed tomography (CT) scanning technique or ≥ 1 cm in the largest dimension by spiral CT scanning (per RECIST criteria); or if, in the Principal Investigator's opinion, evaluable disease can be reliably and consistently followed, the patient may be eligible upon approval by the Onyx Therapeutics, Inc., Medical Monitor.
* Demographic

  * Males and females ≥ 18 years of age
  * Life expectancy of more than three months
  * Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Laboratory

  * Adequate hepatic function, with bilirubin ≤ 1.5 times the upper limit of normal (ULN), and alanine aminotransferase (ALT) ≤ 3 times ULN or ≤ 5 times ULN in the presence of hepatic tumor involvement
  * Absolute neutrophil count (ANC) ≥ 1500/mm3, hemoglobin ≥ 8 g/dL, and platelet count ≥ 100,000/ mm3

    1. Screening platelet count must be independent of platelet transfusions for at least one week
    2. Screening ANC must be independent of granulocyte- and granulocyte/macrophage colony stimulating factor (G-CSF and GM-CSF) support for at least one week and of pegylated G-CSF for at least two weeks
    3. Patients may receive red blood cell (RBC) transfusions or receive supportive care with erythropoietin or darbepoetin in accordance with institutional guidelines
  * Calculated or measured creatinine clearance of ≥ 30 mL/min; calculation using a generally accepted formula such as that of Cockcroft and Gault: CrCl = [(140 - Age) × Mass (kg) / (72 × Creatinine mg/dL)], multiply by 0.85 if female
* Ethical / Other

  * Written informed consent in accordance with federal, local, and institutional guidelines
  * Female patients of childbearing potential must have a negative serum or urine pregnancy test within three days of the first dose and agree to use dual methods of contraception during the study and for one month following the last dose of study drug. Post-menopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from these requirements. Male patients must use an effective barrier method of contraception during the study and for one month following the last dose if sexually active with a female of childbearing potential.

Exclusion Criteria:

* Disease Related

  * Chemotherapy with approved or investigational anticancer therapeutics, including steroid therapy, within four weeks prior to first dose of Oprozomib or six weeks for antibody therapy
  * Radiation therapy or immunotherapy within three weeks prior to first dose; localized radiation therapy within one week prior to first dose Patients with brain metastases (patients with prior brain metastases are permitted, but must have completed treatment and have no evidence of active CNS disease for at least three months prior to first dose)
  * Prior treatment with a proteasome inhibitor
* Concurrent Conditions

  * Major surgery within three weeks prior to first dose
  * Congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, or conduction abnormalities. Conduction system abnormalities not clinically warranting intervention are allowed.
  * Myocardial infarction within three months prior to first dose
  * Active infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
  * HIV infection (HIV seropositive)
  * Active hepatitis A, B, or C infection
  * Peripheral neuropathy of Grade ≥ 3 or Grade 2 with pain at the time of the first dose
  * Patients with pleural effusions requiring repeat thoracentesis or ascites requiring repeat paracentesis
  * Prior Oprozomib therapy
  * Hypersensitivity to Oprozomib or any of its components
* Ethical / Other

  * Female patients who are pregnant or lactating
  * Psychiatric or medical conditions that in the opinion of the Investigator could interfere with treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD) | 31 months
  * To evaluate the safety and tolerability of Oprozomib in patients with advanced refractory or recurrent solid tumors including determination of its Dose Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD)
  * To determine the pharmacokinetics (PK) of Oprozomib

SECONDARY OUTCOMES:
Overall response rate (ORR), duration of responses (DOR), progression-free survival (PFS), and time to progression (TTP) | 31 months
  * To explore the anti-tumor activity of Oprozomib in this patient population including the overall response rate (ORR), the duration of responses (DOR), the progression-free survival (PFS) and time to progression (TTP)
  * To define the pharmacodynamics (PDn) of Oprozomib.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Oncology Research Associates, Scottsdale, Arizona
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas